CLINICAL TRIAL: NCT04913584
Title: Online Peer-Delivered Group Cognitive Behavioural Therapy for Postpartum Depression: A Randomized Controlled Trial
Brief Title: Peer Administered Online CBT for PPD
Acronym: PL-OCBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Kids Can Fly (Unknown)
Responsible Party: Principal Investigator, Ryan Van Lieshout, MD, PhD, Assistant Professor, Department of Psychiatry and Behavioural Neurosciences, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PL OCBT
Record Dates: First submitted 2021-05-29; First posted 2021-06-04 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Postpartum Depression
Keywords: Postpartum depression; CBT; Lay Peer; Online therapy
MeSH Terms: conditions — Depression, Postpartum | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Intervention (Experimental): Online Group CBT for PPD. Women in the treatment group will attend an online 9-week group Cognitive Behavioural Therapy intervention for PPD. This intervention was developed at the Women's Health Concerns Clinic (WHCC) at St. Joseph's Healthcare Hamilton and designed to be brief, simple, and applicable to women in community settings. It consists of 9 weekly 2-hour sessions where core CBT skills are learned and practiced, and a new psychoeducational topic is introduced and discussed by women each week. The CBT intervention will be delivered by eight lay-peers.
  Interventions: Behavioral: Cognitive Behavioural Therapy
- Wait-List Controls (Experimental): Online Group CBT for PPD 9 weeks after enrollment. The women in this arm of the study will receive the same Cognitive Behavioural Therapy intervention as in the immediate intervention arm, however, they will begin the CBT group 9 weeks after enrolling in the study.
  Interventions: Behavioral: Cognitive Behavioural Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioural Therapy — Cognitive Behavioral Therapy 9 weekly 2-hour online group CBT sessions delivered by trained lay peers.

SUMMARY:
Postpartum depression (PPD) affects up to one in five of women and has profound effects on mothers and their infants. Unfortunately, fewer than 15% of women with PPD receive evidence-based care. This is at least partly due to significant difficulties faced by women in accessing psychotherapies, their preferred treatment for PPD. Around the world, there is a significant lack of healthcare professionals trained to deliver CBT. This study will utilize a randomized controlled trial design (with wait-list controls) and recruit 174 participants to determine if women with a past history of PPD (i.e., lay peers) can be trained to deliver effective group CBT online to women currently struggling with PPD. If peers can be trained to provide effective CBT, more women would receive treatment and the burden of PPD on women, families, and the healthcare system would be significantly reduced.

DETAILED DESCRIPTION:
Postpartum depression (PPD) affects up to 20% of women and has profound effects on mothers and their infants. Indeed, the cost of one case of PPD is estimated to exceed $150,000. Unfortunately, fewer than 15% of women with PPD receive evidence-based care and this is at least partly due to difficulties accessing treatment, particularly those that are most preferred (e.g., psychotherapy).

Clinical practice guidelines recommend that the majority of women with PPD receive psychotherapy (e.g., cognitive behavioural therapy (CBT)) as a 1st-line treatment and that screening only occur in settings where CBT is readily available. In order to increase access to treatment, screening efforts have been undertaken by public health units across Canada. This is despite recommendations that this only be conducted in the setting of timely access to evidence-based psychotherapies (e.g., CBT). The purpose of this study is to apply task shifting to the treatment of PPD by determining if women with a past history of PPD (i.e., lay peers) living in the community can be trained to deliver effective group CBT to women with current PPD.

A group CBT intervention for PPD has been developed and validated as well as a training program that pilot data suggests is capable of successfully training public health nurses with little background psychiatric training. This intervention is brief, effective, and generalizable to women with PPD in the community. Peer administered interventions (PAIs), those delivered by recovered former patients are increasingly recognized as potentially effective alternatives to traditional mental health care services. In addition, psychotherapy delivered online has been recognized as a delivery method that results in successful expression and interpretation of emotions, decreased inhibition and reluctance to disclose personal information and a strong therapeutic alliance between patients and providers. Online psychotherapy also has satisfaction ratings that are comparable to traditional in-person psychotherapy.

Eight lay peers will be trained to deliver our 9-week group CBT treatment. 174 women will be recruited and using a randomized controlled trial design (with wait-list controls), it will be determined if lay peers can deliver effective group CBT for PPD.

If peers can be trained to provide effective CBT online, more women would receive treatment and the burden of PPD on women, families, and the healthcare system would be significantly reduced. Providing women with PPD with CBT skills at this crucial stage in life also has the capacity to prevent future depressive relapse with significant benefits for patients, families, employers, and the healthcare system.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* Understand and speak English (so that they can participate in the CBT group and complete study measures)
* Have an EPDS score >10
* Be within 12 months of delivering an infant
* Live within a 2-hour radius of the Brant Region.

Exclusion Criteria:

* Bipolar disorder
* Current psychotic disorder
* Substance use disorder
* Alcohol use disorder
* Antisocial or borderline personality disorder

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2022-02-22 (Actual); Study Completion 2022-02-22 (Actual)

PRIMARY OUTCOMES:
Edinburgh Postnatal Depression Scale | 6 months
  The EPDS will be used to assess maternal depression. A score of >10 is consistent with probable PPD and changes in scores >4 are indicative of clinically significant improvement.

SECONDARY OUTCOMES:
Postpartum Bonding Questionnaire | 6 months
  Used to detect disorders of the mother-infant relationship. Higher scores indicate more impaired bonding.
Social Provisions Scale | 6 months
  Used to measure the degree to which mothers' social relationships provide support. Higher scores indicate higher levels of social support.
Canadian Community Health Survey Maternal Healthcare Utilization | 6 months
  Adopted from the Canadian Community Health Survey to Track use of healthcare services by mothers and their infant.
Adult Adolescent Parenting Inventory | 6 months
  Used to assess the parenting and child rearing attitudes of parents. Higher scores indicate lower risk parenting.
EuroQol-5D | 6 months
  Used to measure health-related quality of life. Higher scores indicate more severe or frequent problems.
Generalized Anxiety Disorder-7 | 6 months
  Used to assess generalized anxiety disorder, the most common comorbidity of postpartum depression. Higher scores indicate more severe generalized anxiety disorder symptoms.
Mini International Neuropsychiatric Interview - Current Major Depressive Disorder | 6 months
  Used to assess maternal depression.
Parenting Stress Index (Short-Form) | 6 months
  Used to measure stress in parent-child relationships. Higher scores indicate higher levels of stress.
Infant Behavior Questionnaire-Revised | 6 months
  Used to measure infant temperament. Higher scores indicate greater levels of the specific temperament dimension.
Ages and Stages Questionnaire | 6 months
  Used to measure communication and motor development in children. Higher scores indicate more positive outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Van Lieshout, MD, PhD, Principal Investigator — McMaster University
Locations (1):
- Kids Can Fly, Brantford, Ontario, Canada